CLINICAL TRIAL: NCT02390544
Title: Melphalan Pharmacokinetics in Children Undergoing Hematopoietic Stem Cell Transplantation: A Pilot Study
Brief Title: A Pharmacokinetic Study of Melphalan in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-5123
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: children; bone marrow transplant; pharmacokinetics
MeSH Terms: interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melphalan in Patients Receiving HSCT (Experimental): The investigators will recruit approximately 30 patients who are scheduled to undergo allogeneic transplant with reduced intensity conditioning that includes melphalan. Approximately 10 patients who will receive melphalan as part of their conditioning regimen for an autologous transplant will also be recruited.
  A test dose of melphalan will be administered prior to the start of the HSCT preparative regimen. The test dose will equal 10% of the standard dose. Blood samples will be drawn for pharmacokinetic measurement prior to and after the administration of the test dose and again around the full standard dose of melphalan. Urine samples will also be collected around the test dose and full standard dose of melphalan to measure markers of kidney injury.
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Melphalan — Melphalan is a bifunctional alkylating agent that inhibits DNA and RNA synthesis, cross-links strands of DNA and acts on both resting and rapidly dividing cells including tumor cells. It is administered intravenously.
  Other Names: Alkeran

SUMMARY:
The purpose of this study is to examine the pharmacokinetics (PK) of melphalan in children undergoing hematopoietic stem cell transplantation (HSCT). Melphalan is an important component of HSCT preparative regimens, but can be associated with significant toxicity. PK data is a powerful clinical tool that, when used to develop individualized treatment plans for a specific patient, may ultimately increase the likelihood of selecting the right dose for the right patient and/or of reducing the number of adverse drug events. The investigators' goal is to establish baseline pediatric melphalan PK data. These data may be used for patient specific dosing of melphalan in the future to minimize toxicity and improve transplant outcomes.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) continues to be the only curative therapy for patients with many hematological diseases. The adverse effects associated with chemotherapy agents used as part of HSCT preparative regimens are not insignificant and can be life threatening at times. The investigators' central hypothesis is that increased systemic exposure to melphalan due to variation in PK in younger children leads to increased toxicity seen in them. Although the PK of melphalan has been studied in animal models and in adult patients, limited data exists in pediatric patients especially those undergoing allogeneic HSCT. The objective of this study is to describe the pharmacokinetics of melphalan in children undergoing hematopoietic stem cell transplantation. Up to forty patients who are scheduled to receive melphalan as part of their preparative regimen will be enrolled. Prior to the start of the preparative regimen, study participants will receive a test dose of melphalan (10% of the standard dose). Blood samples will be collected at specific time points prior to and after the administration of the test dose and again around the full standard dose of melphalan. This study will establish that a novel method (dry blood spot assay) of determining PK of melphalan can be utilized in the clinical setting. Additionally, urine samples will be collected to measure markers of kidney injury, which will help correlate melphalan exposure with toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either allogeneic RIC HSCT, or autologous transplant containing melphalan as part of the preparative regimen at CCHMC will be included.

Exclusion Criteria:

* Failure to sign informed consent, or inability to undergo informed consent process.
* It is not medically advisable to obtain the specimens necessary for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of melphalan in children undergoing HSCT | Prior to the melphalan infusion, and then approximately 5 min, 15 min, 30 min, 45 min, 60 min, 2, 2.5, 4, and 6 hours after the end of the melphalan infusion.
  Blood samples will be collected at the above time points around the test dose of melphalan and again around the standard full dose of melphalan. AUC will be used to characterize the pharmacokinetics of melphalan.

SECONDARY OUTCOMES:
Perform measurement of acute kidney injury marker, KIM-1 | Prior to the melphalan infusion and approximately 8 hours and 24 hours following the end of melphalan infusion.
  Urine samples will be collected at the above time points around the test dose of melphalan and again around the standard full dose of melphalan for measurement of KIM-1.
Perform measurement of acute kidney injury marker, NGAL | Prior to the melphalan infusion and approximately 8 hours and 24 hours following the end of melphalan infusion.
  Urine samples will be collected at the above time points around the test dose of melphalan and again around the standard full dose of melphalan for measurement of NGAL.

CONTACTS AND LOCATIONS:
Overall Officials: Sharat Chandra, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Parinda Mehta, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States